CLINICAL TRIAL: NCT06393634
Title: Comparing Direct and Indirect Detection Methods Following Multiple Routes of Testosterone administration-an Anti-doping Perspective
Brief Title: Comparing Direct and Indirect Detection Methods of Multiple Routes of Testosterone Administration
Acronym: T esters
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sports Medicine Research and Testing Laboratory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMRTL.2024.01
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Testosterone; Testosterone Propionate; testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: Three groups in phase one and two groups in phase two, randomized by a computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone group one (Active Comparator): The participant will receive a single injection of one of three types of testosterone in phase one.
  In phase two the participant will receive two weeks of either a daily skin cream or a twice-daily pill to swallow.
  Interventions: Drug: Testosterone injection; Drug: Testosterone gel
- Testosterone group two (Active Comparator): The participant will receive a single injection of one of three types of testosterone in phase one.
  In phase two the participant will receive two weeks of either a daily skin cream or a twice-daily pill to swallow.
  Interventions: Drug: Testosterone injection; Drug: Testosterone Oral

INTERVENTIONS:
Drug: Testosterone injection — A single injection of testosterone
  Other Names: testosterone cipionate, enanthate,or propionate
Drug: Testosterone gel — A daily dose of testosterone gel
  Other Names: testosterone transdermal
  Arms: Testosterone group one
Drug: Testosterone Oral — A twice-daily pill of testosterone pill to swallow
  Other Names: testosterone undecanoate
  Arms: Testosterone group two

SUMMARY:
Testosterone abuse is extremely prevalent in athletes globally and especially in the United States professional sporting leagues

DETAILED DESCRIPTION:
Because human bodies make testosterone naturally, it can be difficult to determine whether the testosterone in your body is natural or if it came from administering testosterone. Currently, testosterone abuse by athletes is detected by anti-doping laboratories in urine samples and use can also be inferred by testing blood samples. As a pharmaceutical preparation, testosterone is available to administer to your body in different ways. However, due to lack of controlled data on the various preparations of testosterone administrations related to the anti-doping field, this study id designed to look at five different testosterone preparations delivered three different ways and how they compare to each other in terms of anti-doping detection and how long they will be in circulation in your body.

ELIGIBILITY:
Inclusion Criteria:

* HEALTHY MALE ADULTS, AGED 18-60 YEARS

Exclusion Criteria:

* Individuals currently enrolled in a registered testing pool for anti-doping purposes
* Unwilling to provide urine or blood samples
* Individuals who are not actively exercising
* Individuals who show a high risk of heart attack or cardiovascular disease as defined by a physician
* Individuals that have an elevated baseline hematocrit as determined by the PI
* Individuals who are diabetic or are currently taking diabetic medications.
* Individuals that have donated blood (approximately 500 mL) in the past 8 weeks
* Individuals with severe acne
* Individuals with a history of cancer, cardiac, renal or hepatic disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Detection windows of testosterone administered via injection, oral and skin cream. | 12 weeks
  Changes in urinary testosterone/epitestosterone ratio after administration of testosterone in injection, oral and cream
Changes in serum concentration of testosterone | 12 weeks
  Changes in serum concentrations of testosterone in injection, oral and cream administration of testosterone
Changes in serum concentration of androstenedione | 12 weeks
  Changes in serum concentrations of androstenedione in injection, oral and cream administration of testosterone
Changes in serum concentration of luteinizing hormone | 12 weeks
  Changes in serum concentrations of luteinizing hormone after injection, oral and cream administration of testosterone

SECONDARY OUTCOMES:
Direct detection of testosterone esters | 12 weeks
  Direct detection of testosterone esters

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Miller, PhD, Study Director — Sports Medicine Research and Testing Laboratory
Locations (1):
- Sports Medicine Research and Testing Laboratory, South Jordan, Utah, United States

IPD SHARING:
Plan to Share IPD: No